CLINICAL TRIAL: NCT01048645
Title: Randomized Phase II Trial: Effect of All-trans Retinoic Acid With Chemotherapy Based in Paclitaxel and Cisplatin as First Line Treatment of Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Effect of All-trans Retinoic Acid With Chemotherapy Based in Paclitaxel and Cisplatin as First Line Treatment of Patients With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Cancerología (Other Government)
Collaborators: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Oscar Arrieta, Instituto Nacional de Cancerología
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICC/302/07
Record Dates: First submitted 2009-12-30; First posted 2010-01-13 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: All-trans retinoic acid; non-small cell lung cancer; retinoic acid receptor beta; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- P/PC arm (Placebo Comparator): Patients were assigned to receive placebo (P/PC) 1 week prior to treatment until completing two cycles
  Interventions: Other: PLACEBO
- RA/PC arm (Experimental): Patients were assigned to receive ATRA 20 mg/m2/day (RA/PC) 1 week prior to treatment until completing two cycles
  Interventions: Drug: ATRA

INTERVENTIONS:
Drug: ATRA — Patients were assigned to receive ATRA 20 mg/m2/day (RA/PC) 1 week prior to treatment until completing two courses of chemotherapy based on paclitaxel and cisplatin
  Arms: RA/PC arm
Other: PLACEBO — Patients were randomized to receive or placebo (P/PC) 1 week prior to treatment until completing two courses of chemotherapy based on paclitaxel and cisplatin
  Arms: P/PC arm

SUMMARY:
Purpose:

This randomized phase II trial evaluated whether the combination of cisplatin and paclitaxel plus All-trans retinoic acid (ATRA) increases Response rate (RR) and Progression-free survival (PFS) in patients with advanced Non-small cell lung cancer (NSCLC) with an acceptable toxicity profile and its association with the expression of Retinoic acid receptor beta 2 (RAR-beta2) as a response biomarker.

Patients and Methods:

Patients with stage IIIB and IV NSCLC were included to receive Paclitaxel and Cisplatin (PC). Patients were randomized to receive ATRA 20 mg/m2/day (RA/PC) or placebo (P/PC) 1 week prior to treatment until completing two cycles. RAR-beta2 expression was analyzed by Immunohistochemistry (IHC) and RT-PCR in tumor and adjacent lung tissue.

DETAILED DESCRIPTION:
Purpose:

This randomized phase II trial evaluated whether the combination of cisplatin and paclitaxel plus All-trans retinoic acid (ATRA) increases Response rate (RR) and Progression-free survival (PFS) in patients with advanced Non-small cell lung cancer (NSCLC) with an acceptable toxicity profile and its association with the expression of Retinoic acid receptor beta 2 (RAR-beta2 ) as a response biomarker.

Patients and Methods:

Patients with stage IIIB and IV NSCLC were included to receive Paclitaxel and Cisplatin (PC). Patients were randomized to receive ATRA 20 mg/m2/day (RA/PC) or placebo (P/PC) 1 week prior to treatment until completing two cycles. RAR-beta2 expression was analyzed by Immunohistochemistry (IHC) and RT-PCR in tumor and adjacent lung tissue.

ELIGIBILITY:
Inclusion Criteria:

* Stage III B and IV NSCLC
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* No prior cytotoxic chemotherapy for NSCLC
* Age ≥18 years, adequate laboratory measurements
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST)
* Life expectancy of >12 weeks.

Exclusion Criteria:

* Patients who had received prior chemotherapy
* Patients with other comorbid conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2007-09; Primary Completion 2008-12 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The primary end-point was Response rate (RR) and Progression-free survival (PFS), as well as identifying whether expression of RAR-beta2 is a response biomarker. | 2 years

SECONDARY OUTCOMES:
Evaluate the efficiency and safety of low doses of ATRA in patients with advanced NSCLC who receive first-line CT. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Arrieta, M.D., Principal Investigator — National Institute of Cancerología
Locations (1):
- National Institute of Cancerología, Mexico City, Mexico City, Mexico